CLINICAL TRIAL: NCT01187264
Title: Efficacy and Safety of Methotrexate in 2 Fixed Doses of 10mg or 25mg Orally Once Weekly in Patients With Severe Plaque Type Psoriasis: a Prospective, Randomized, Double Blind, Dose Ranging Study
Brief Title: Dose Ranging Study to Compare the Efficacy and Safety of Methotrexate in Plaque Type Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr C Vijay Krishna, postgraduate institute of medical education and research
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7557/PG/2Trg/07
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2009-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methotrexate 10 mg (Active Comparator): oral methotrexate 10 mg once weekly
  Interventions: Drug: Methotrexate
- methotrexate 25mg (Active Comparator): oral methotrexate 25 mg once weekly
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — once weekly for a total duration of 12 weeks or earlier till patient achieves PASI 75

SUMMARY:
In this study the investigators intend to compare the efficacy and safety of two fixed doses of once weekly oral methotrexate in a prospective randomized double blind manner in patients with severe plaque type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plaque-type psoriasis having more than 10% body surface area involvement (severe psoriasis).20
* Patients of either sex with age between 18-65 years.
* Females who were postmenopausal or tubectomised or have completed their family size and are willing to maintain contraception 1 month before, during and 1 month after completion/stopping of treatment and negative pregnancy test 2 weeks before starting of treatment and at day 2 or 3 of a normal menstrual cycle.
* Males who were willing to maintain contraception during and 3 months after completion/stopping of treatment.

Exclusion Criteria:

* Pregnant or lactating women.
* Any abnormalities in renal function, cardiovascular disease, respiratory disease or neuropsychiatric illness.
* Significant abnormalities in liver function (serum bilirubin, AST, ALT, and ALP >1.5 times the upper limit of normal), viral hepatitis or cirrhosis.
* history of excessive alcohol consumption.
* Severe anemia, leucopenia or thrombocytopenia.
* Active infectious disease or immune system deficiency including AIDS.
* history of intolerance/hypersensitivity to methotrexate.
* history of phototherapy in past 6 months.
* Patients who had received any systemic treatment for psoriasis in the past 4 weeks and topical treatment in the past 2 weeks.
* Body mass index (BMI) > 30 kg/m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
change in Psoriasis Area and Severity Index (PASI) score between two groups from baseline to 12 weeks | 12 weeks

SECONDARY OUTCOMES:
time to achieve PASI 75 | 12 weeks or earlier
number of patients achieving PASI 90 and 100 | 12 weeks or earlier

CONTACTS AND LOCATIONS:
Overall Officials: C V KRISHNA, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; SUNIL DOGRA, MD, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, U.T, India